CLINICAL TRIAL: NCT06528756
Title: Calciying Tendinopathy of the Rotator Cuff: Barbotage Vs Shock Waves
Acronym: BOTCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Javier Muñoz Paz, Medicine ( Principal Investigator), Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOTCH
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Tendinopathy Rotator Cuff; Calcific Tendinitis; High-Energy Shock Waves; Barbotage; Pain, Shoulder
Keywords: Tendinopathy Rotator Cuff; Calcific Tendinitis; High-Energy Shock Waves; Barbotage; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Prospective block-randomized experimental longitudinal analytical clinical trial
  Patients will be stratified into two arms according to the Bianchi Martinoli classification (I or II/III) and will subsequently be included in groups based on the treatment received, US-PICT or ESWT . The decision to treat with one or another therapy will be made randomly 1:1, based on the treatment assigned to the previous patient. An initial consultation and 3 reviews (1 month, 3 months and 6 months) will be carried out after completing the therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type I calcifications (Active Comparator): Type I calcifications according to the Bianchi Martinoli classification
  Interventions: Procedure: shockwave therapy; Procedure: Barbotage
- Type II/III calcifications (Active Comparator): Type II/III calcifications according to the Bianchi Martinoli classification
  Interventions: Procedure: shockwave therapy; Procedure: Barbotage

INTERVENTIONS:
Procedure: shockwave therapy — ESWT, these will be given using a 15 mm transmitter in mode continuous with pressure at 3 bar, frequency 12Hz and 3000 impacts. The number of sessions will be between 4 - 8 depending on the patient's clinic with a break between sessions of 5 to 10 days.
  Other Names: ESWT
Procedure: Barbotage — US-PICT will be carried out with 1 session in which the following actions will be carried out:
  * First, a suprascapular nerve block will be performed with a corticosteroid and anesthetic (3 ml of bupivacaine) in an ultrasound-guided manner.
  * The calcification will then be infiltrated with 5 ml local lidocaine and preloaded physiological saline solution in an ultrasound-guided manner.
  * Finally, repeated suctions will be performed with physiological saline solution to extract calcium in an ultrasound-guided way.
  Other Names: US-PICT

SUMMARY:
The objective of this block randomized prospective experimental longitudinal analytical clinical trial is to compare the mean differences in Visual analgesic scale (VAS) at 1 month, 3 months and 6 months depending on the treatment received, ultrasound-guided barbotage (US-PICT) or shock waves (ESWT), in patients with calcifying tendinopathies according to the lesion based on the Bianchi Martinolli classification, as well as to know if there are variations in functionality with the Latinen test, joint balance, patient global improvement impression scale (PGI-I), global improvement impression scale (CGI - GI).

For this purpose, patients between 30 and 60 years old, with chronic shoulder pain for more than 3 months due only to calcifying tendinopathies who have not received these previous treatments will be selected.

The main question to be answered is:

Do patients with calcifying tendinopathies of the shoulder, in its different degrees, who have received as treatment barbottage, obtain the same VAS differences at 1 month, 3 month and 6 month as patients who received as treatment shock waves in the population?

Patients will be sorted into two arms according to the Bianchi Martinoli classification (I or II/ III) and subsequently included in groups according to the treatment received. The decision to treat with one or the other therapy will be made randomly 1:1, depending on the treatment assigned to the previous patient. An initial consultation and 3 revisions (1 month, 3 months and 6 months) will be performed after the end of therapy.

The following variables will be collected VAS, Lattinen test, joint balances (ROM) (flexion, abduction and external and internal rotation), PGI-I, CGI - GI.

DETAILED DESCRIPTION:
Shoulder pain is a very common health issue among adults, being 8% due to calcifying tendinopathies of the shoulder (CT). The evolutionary process of this lesion can be classified according to Bianchi Martinoli as I: hard, II: semi-soft and III: soft due to their ultrasound appearance.

In 50% of cases, with first-line treatments such as kinesitherapy and taking anti-inflammatories, they resolve spontaneously. However, in the remaining 50% they become chronic, requiring other lines of treatment such as shock waves (ESWT) or ultrasound-guided barbotage (US-PICT).

Starting hypothesis:

Patients with CT, in its different degrees, who have received barbottage as treatment, obtain the same VAS differences at 1 month, 3 months and 6 months as patients who received ESWT as treatment in the population.

Main objective:

* The main objective is to compare the mean differences in VAS at 1 month, 3 months and 6 months according to the treatment received, barbotage or ESWT in patients with CT according to the evolutionary stage of the lesion based on the Bianchi Martinolli classification.

Secondary objectives:

* To know if there are variations in functionality with the Latinen test, joint balance (ROM), PGI and CGI.
* To protocolize an attitude towards this type of pathology.
* To favor the use of hospital resources.

We propose to conduct a block randomized prospective experimental longitudinal analytical block randomized clinical trial. For this purpose, patients aged between 30 - 60 years, with chronic shoulder pain for more than 3 months due only to calcifying tendinopathies will be selected.

The protocol carried out was as follows:

1. st Phase : in this first phase, patients will be collected according to the criteria set out above for a period of 12 months. During this time, the patients will be explained the two possible treatments to be received and after signing the appropriate informed consent, they will be divided into groups according to treatment (ESWT vs US-PICT) stratifying according to the Bianchi Martinolli classification: (I or II/IIII). The decision for each treatment will be made randomly, dividing the patients in a 1:1 ratio according to whether they attend the initial consultation and the previous patient has received one or the other treatment.
2. nd Phase: Subsequently, 3 revisions will be performed. One at 1 month, 3 months and another one at 6 months after the end of the therapy.
3. rd Phase: The information collected will be synthesized and entered into the SPSS V.21 program to obtain results.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 30 - 60 years.
* Omoalgia lasting more than 3 months.
* Radiographic and ultrasound visualization in both planes of calcification.
* Sizes > 5 millimeters (mm).

Exclusion criteria:

* Patients who do not meet inclusion criteria.
* Presence of another obvious cause of pain (joint degeneration, capsulitis, rotator cuff tendon tears...)
* Previously received barbotage or shock waves.
* Contraindication of therapies: infection, allergies to medications, cancer...

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-11-23 (Actual); Study Completion 2025-11-23 (Actual)

PRIMARY OUTCOMES:
Visual analgesic pain scale (VAS) | 6 months
  The VAS will be measured in the initial consultation and at 1, 3 and 6 months after the intervention and a new variable "VAS Difference" (DifVAS) will be created for each corresponding VAS level in the review consultations.

SECONDARY OUTCOMES:
Latineen test | 6 months
  The Latineen test is a widely used tool for pain evaluation. Initial, at 1, 3 and 6 months of each variable. It contains five subscales that score from 0 to 4:
  1. Pain intensity. 2. Frequency of pain. 3. Consumption of painkillers. 4. Degree of disability. 5. Hours of sleep.
Patient Global Patient Improvement Impression Scale (PGI-I) | 6 months
  The PGI-I consists of a single question that asks the patient to classify the relief obtained with the treatment according to a 7-point Likert scale: "much better"; "much better"; "a little better"; "no change"; "a little worse"; "much worse"; "much worse".
Global CGI - GI Impression of Global Improvement Scale (CGI - GI) | 6 months
  The CGI-Improvement (CGI-I) , the physician compares the patient's initial clinical condition with the current condition: "Compared to the patient's condition at the time of admission to the project [prior to the start of medication], this patient's condition is: 1=much better since the start of treatment; 2=much improved; 3=minimally improved; 4=no change since baseline (the start of treatment); 5=minimally worse; 6=much worse; 7=much worse since the start of treatment."
Shoulder joint balances (ROM) | 6 months
  Flexion, abduction and external and internal rotation (º) measured with goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Muñoz Paz, Medicine, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvie P, Pollard TC, Carr AJ. Calcific tendinitis: natural history and association with endocrine disorders. J Shoulder Elbow Surg. 2007 Mar-Apr;16(2):169-73. doi: 10.1016/j.jse.2006.06.007. Epub 2006 Dec 22. PMID 17188907
- [Background] Ejnisman B, Andreoli CV, Monteiro GC, Pocchini Ade C, Cohen C, Tortato S, Franklin MM, Machado AB, Cohen M. CALCIFYING TENDINOPATHY: A LOCAL OR A SYSTEMIC CONDITION? Rev Bras Ortop. 2015 Dec 8;47(4):479-82. doi: 10.1016/S2255-4971(15)30132-4. eCollection 2012 Jul-Aug. PMID 27047854
- [Background] Chianca V, Albano D, Messina C, Midiri F, Mauri G, Aliprandi A, Catapano M, Pescatori LC, Monaco CG, Gitto S, Pisani Mainini A, Corazza A, Rapisarda S, Pozzi G, Barile A, Masciocchi C, Sconfienza LM. Rotator cuff calcific tendinopathy: from diagnosis to treatment. Acta Biomed. 2018 Jan 19;89(1-S):186-196. doi: 10.23750/abm.v89i1-S.7022. PMID 29350647
- [Background] Gerdesmeyer L, Wagenpfeil S, Haake M, Maier M, Loew M, Wortler K, Lampe R, Seil R, Handle G, Gassel S, Rompe JD. Extracorporeal shock wave therapy for the treatment of chronic calcifying tendonitis of the rotator cuff: a randomized controlled trial. JAMA. 2003 Nov 19;290(19):2573-80. doi: 10.1001/jama.290.19.2573. PMID 14625334
- [Background] Ramon S, Espanol A, Yebra M, Morillas JM, Unzurrunzaga R, Freitag K, Gomez S, Aranzabal JR. [Current evidences in shockwave treatment. SETOC (Spanish Society of Shockwave Treatment) recommendations]. Rehabilitacion (Madr). 2021 Oct-Dec;55(4):291-300. doi: 10.1016/j.rh.2021.02.002. Epub 2021 Mar 17. Spanish. PMID 33743978
- [Background] Sanchez Lite I, Toribio Calvo B, Osorio Aira S, Romera de Blas C, Andres Garcia N. Treatment of calcific tendinopathy of the rotator cuff with ultrasound-guided puncture and aspiration. Radiologia (Engl Ed). 2021 Aug 26:S0033-8338(21)00124-7. doi: 10.1016/j.rx.2021.07.005. Online ahead of print. English, Spanish. PMID 34456048
- [Background] García A. Nicolás, Rosales L. Julio, Verdugo P. Marco Antonio. Tendinopatía cálcica: Etiopatogenia y evaluación por imágenes. Rev. chil. radiol. 2020 Jun; 26(2): 52-61.
- [Background] González-Escalada J. R., Camba A., Muriel C., Rodríguez M., Contreras D., Barutell C. de. Validación del índice de Lattinen para la evaluación del paciente con dolor crónico. Rev. Soc. Esp. 2012 Ago; 19(4): 181-188.
- [Background] Estenne M, Yernault JC. The mechanism of CO2 retention in cardiac pulmonary edema. Chest. 1984 Dec;86(6):936-8. doi: 10.1378/chest.86.6.936. PMID 6437753
- [Background] Bianchi S, Martinoli C. Extremidad superior. In: Ecografia Musculoesquelética; Baert A.L, Knauth M, Sartor K, editores; MARBAN; 2011; pp 159-294.
- [Result] Berrigan W, Olufade O, Negron G, Easley K, Sussman WI. Calcific Tendinopathy of the Shoulder: A Retrospective Comparison of Traditional Barbotage Versus Percutaneous Ultrasonic Barbotage. Clin J Sport Med. 2022 Sep 1;32(5):458-466. doi: 10.1097/JSM.0000000000001039. Epub 2022 Apr 22. PMID 35533134
- [Result] Louwerens JK, Sierevelt IN, van Noort A, van den Bekerom MP. Evidence for minimally invasive therapies in the management of chronic calcific tendinopathy of the rotator cuff: a systematic review and meta-analysis. J Shoulder Elbow Surg. 2014 Aug;23(8):1240-9. doi: 10.1016/j.jse.2014.02.002. Epub 2014 Apr 26. PMID 24774621
- [Result] Kim YS, Lee HJ, Kim YV, Kong CG. Which method is more effective in treatment of calcific tendinitis in the shoulder? Prospective randomized comparison between ultrasound-guided needling and extracorporeal shock wave therapy. J Shoulder Elbow Surg. 2014 Nov;23(11):1640-6. doi: 10.1016/j.jse.2014.06.036. Epub 2014 Sep 12. PMID 25219475
- See also: Calcific tendinopathy of the shoulder - Up to date — https://www.uptodate.com/contents/calcific-tendinopathy-of-the-shoulder/print?source=mostViewed_widget
- See also: Unreferenced articles from Pubmed — https://drive.google.com/drive/folders/1SGNjNZ4Om8G7NH-uxv9J63CAn4daY4Ou?usp=sharing

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT06528756/Prot_SAP_002.pdf
  • Informed Consent Form (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT06528756/ICF_001.pdf